CLINICAL TRIAL: NCT06674538
Title: Phase 1, Open Label Clinical Trial to Treat Stage IV Cancer Patients With Multiple Patient-specific Mutated Cell Surface Proteins With Chimeric Antibodies
Brief Title: Clinical Trial to Treat Stage IV Cancer Patients
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Moonshot Antibodies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Moonshot protocol #2024-01
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Soft Tissue Cancer
Keywords: Stage IV cancer; patient-specific mutated cell surface proteins; chimeric antibodies
MeSH Terms: conditions — Sarcoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Treatment with multiple patient-specific mutated cell surface proteins with chimeric antibodies
  Interventions: Drug: Moonshot antibodies

INTERVENTIONS:
Drug: Moonshot antibodies — Chimeric antibodies

SUMMARY:
The purpose of this research is to study the safety and effectiveness of investigational antibodies attacking certain areas on the surface of cancer cells so that the body can kill the cancer cells. The antibodies will be made in a laboratory from cells taken from each subject's tumor so they will be made specifically per subject.

The first step is to take blood and tumor samples so that the laboratory can produce antibodies specific to each subject's tumor. During this process, the study team will identify specific areas on the cancer cells that are not normally present in healthy cells so that the antibodies can find the cancer cells that should be destroyed.

The second step is to deliver the antibodies to each subject through a series of infusions.

DETAILED DESCRIPTION:
This is a Phase I open-label, multicenter study to evaluate the safety and feasibility of treating with chimeric antibodies that target mutated cell surface proteins.

Up to 12 evaluable subjects will be treated at up to 5 study sites. Evaluable subjects are those who receive at least 4 doses of treatment. A maximum of 16 subjects will be enrolled, regardless of the number of treatment doses administered.

After consent is obtained to acquire tumor and normal cells, it will be determined if sufficient archived tumor tissue is available. In the absence of sufficient archived tumor tissue, subjects will undergo biopsy of tumor. The aseptic collection of tumor material will occur in a manner suitable for DNA and RNA extraction and sequencing.

Sequencing for this study will be performed in a laboratory that performs whole exome and RNA sequencing. Quality thresholds will include metrics such as base calling quality, coverage, allelic read percentages, strand bias, and alignment quality.

Upon successful antibody production, the antibodies will be delivered to each subject through a series of infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older who have biopsy proven cancer. The following types of malignancy will be eligible:

   Stage IV cancer of the following types: breast cancer, colon cancer, esophageal cancer, kidney cancer, lung cancer, lymphoma, melanoma, ovarian cancer, pancreatic cancer, bladder, urothelial carcinoma, head and neck cancers, prostate cancer, sarcomas, and stomach cancer.
2. Subjects who have refractory or progressive disease after at least 1 line of systemic treatment or who have declined additional curative standard of care therapy(ies).
3. Subjects willing to consent to obtaining a blood sample and archived tumor tissue for genomic extraction and amplification. If archived tumor tissue is not available, a new biopsy sample will be required. If sequencing was previously completed under Moonshot Antibodies IRB protocol #20233336 or completed on the patient's tumor as part of clinical care, these results and samples may be used and duplicative tumor sequencing will not be necessary.
4. Subjects must have measurable disease as defined per the Response Evaluation Criteria in Solid Tumor (RECIST) at the time of biopsy. Archived tumor must be available or tumor must be accessible for biopsy.
5. Karnofsky Score must be ≥ 60
6. Hematological:

   1. ANC (Absolute neutrophil count) ≥ 1000/µl (unsupported)
   2. Platelets ≥ 100,000/µl (can be transfused)
   3. Hemoglobin > 8 g/dL (can be transfused)
7. Renal: Serum creatinine ≤ 1.5 x upper limit of institutional normal.
8. Adequate liver function must be demonstrated, defined as:

   1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   2. ALT (SGPT) ≤ 3 times upper limit of normal (ULN)
   3. AST (SGOT) ≤ 3 times upper limit of normal (ULN)
9. A negative serum pregnancy test is required for female participants of childbearing potential (≥13 years of age or after onset of menses)
10. Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrel implants (Norplant), or medroxyprogesterone acetate injections (Depo-Provera shots). If none of these can be used, contraceptive foam with a condom is recommended.
11. Informed Consent: All subjects must sign written informed consent.

Exclusion Criteria:

1. Insufficient tumor tissue for genome sequencing.
2. Known human immunodeficiency virus infection.
3. Subjects who have received any cytotoxic treatment within 3 weeks of antibody treatment.
4. Subjects who have received any radiotherapy to the tumor biopsy sample site within the last 14 days (radiation may be included in treatment decision after biopsy).
5. Subjects who have received live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.
6. Subjects who are currently receiving or have received systemic therapeutic corticosteroids ≤2 weeks prior to starting treatment.
7. Subjects receiving any investigational drug concurrently.
8. Subjects with chronic active autoimmune diseases undergoing treatment.
9. Subjects who have had prior organ transplant.
10. Subjects who have developed allergic responses to chimeric antibodies.
11. Subjects with symptomatic known brain metastases < 4 weeks from radiation treatment
12. Subjects with significant (>Grade 2 toxicity) renal, cardiac, pulmonary, hepatic or other organ dysfunction.
13. Subjects with secondary cancers that require systemic treatment.
14. Subjects that are pregnant or breastfeeding.
15. Subjects with uncontrolled serious infections or a life-threatening illness (unrelated to tumor) including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
16. Subjects with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a subject's ability to sign the informed consent, and subject's ability to cooperate and participate in the study
17. Adult subjects lacking capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Frequency of Grade III or greater adverse events | From first dose of treatment through endpoint evaluation at 6 months
  Frequency of Grade III or greater adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Krag, MD, Study Chair — Moonshot Antibodies
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared according to the following: (i) the use of a controlled access approach, using a transparent and robust system to review requests and provide secure data access; (ii) seeking consent for sharing IPD from trial participants in all future clinical trials with adequate assurance that patient privacy and confidentiality can be maintained; and (iii) establishing an approach to resource the sharing of IPD which would include considerations for stakeholders such as trial funders, sponsor organizations and users of IPD.
Time Frame: After data analysis and IND closure. End date is undetermined at this time.
Access Criteria: This is undetermined at this time.
URL: https://moonshotab.com/